CLINICAL TRIAL: NCT04316390
Title: Influence of Hesperidin and Vitamin C on Uric Acid Concentration
Acronym: HesperiDrinC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Collaborators: Hochschule Geisenheim University (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Anja Bosy-Westphal, Prof. Dr. Dr. Anja Bosy-Westphal, University of Kiel
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ABW-2020-OS2
Record Dates: First submitted 2020-03-12; First posted 2020-03-20 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Higher Uric Acid Concentrations (>5,5 mg/dl); Healthy
Keywords: hesperidin; vitamin C; uric acid concentration
MeSH Terms: interventions — Hesperidin; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hesperidin (A) (Experimental): study drink without hesperidin and without vitamin C compared to study drink with hesperidin
  Interventions: Dietary Supplement: Control; Dietary Supplement: Hesperidin
- Hesperidin + Vitamin C (B) (Experimental): study drink with vitamin C compared to study drink with hesperidin and vitamin C
  Interventions: Dietary Supplement: Vitamin C; Dietary Supplement: Hesperidin + Vitamin C

INTERVENTIONS:
Dietary Supplement: Control — study drink (two weeks)
  Arms: Hesperidin (A)
Dietary Supplement: Hesperidin — study drink + Hesperidin 600 mg (two weeks)
  Arms: Hesperidin (A)
Dietary Supplement: Vitamin C — study drink + Vitamin C 250 mg (two weeks)
  Arms: Hesperidin + Vitamin C (B)
Dietary Supplement: Hesperidin + Vitamin C — study drink + Hesperidin 600 mg + Vitamin C 250 mg (two weeks)
  Arms: Hesperidin + Vitamin C (B)

SUMMARY:
Aim of the study is to investigate the impact of hesperidin and/or vitamin C on elevated uric acid concentrations.

DETAILED DESCRIPTION:
Duration of the study is 9 weeks. 1) a washout week, 2) two intervention weeks, 3) four weeks washout period, 4) two intervention weeks.

The study is conducted under free living conditions. During washout weeks consumption of orange juice or citrus fruits or vitamin C containing supplements is restricted.

During intervention weeks 200 mL of study drink is consumed daily. And participants are asked to maintain their normal physical activity and habitual diet. Additional citrus or vitamin C containing beverages are not allowed.

At the beginning and the end of each intervention phase uric acid, insulin sensitivity, blood pressure, pulse wave velocity and bioavailability of hesperidin are assessed.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* higher uric acid concentration (≥5.5 mg/dL)
* Informed written consent

Exclusion Criteria:

* pregnancy
* fructose intolerance
* smoking
* gout or medicated hyperuricemia
* diabetes mellitus
* antidiabetic or cytostatic medication
* weight loss (≥5% in the past 3 months)
* consumption of vitamin C-containing supplements
* parallel participation in a clinical trial
* anemia and / or iron deficiency

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in uric acid serum concentrations | Baseline (pre) and post two weeks of intervention
  measured via uric acid serum concentration (mg/dL)

SECONDARY OUTCOMES:
changes in uric acid excretion | Baseline (pre) and post two weeks of intervention
  measured via uric acid excretion in 24h urine (mg/24h)
changes in pulse wave velocity | Baseline (pre) and post two weeks of intervention
  measured via oscillometric method (m/s)
insulin sensitivity | Baseline (pre) intervention periods
  measured via minimal model from oral glucose tolerance test data using the particular study drink with added glucose to 75 g Glucose / 200 mL

OTHER OUTCOMES:
bioavailability of hesperidin in blood | Baseline (pre) and post two weeks of intervention
  detection of hesperidin metabolites measured via chromatography and following mass spectrometry in serum
bioavailability of hesperidin in urine | Baseline (pre) and post two weeks of intervention
  detection of hesperidin metabolites measured via chromatography and following mass spectrometry in 24h urine

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westphal, Prof, PhD, MD, Principal Investigator — Institute of Human Nutrition, Kiel University
Locations (1):
- Institute of Human Nutrition, Kiel, Germany